CLINICAL TRIAL: NCT00004547
Title: Phase II Trial of Continuous Hyperthermic Peritoneal Perfusion (CHPP) With Cisplatin Plus Early Postoperative Intraperitoneal Paclitaxel and 5-Fluorouracil for Peritoneal Carcinomatosis
Brief Title: Treatment of Peritoneal Cancer With Surgery, Perfused Heated Cisplatin and Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Marybeth Hughes, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 000069; 00-C-0069; NCT00020059 (obsolete NCT alias)
Record Dates: First submitted 2000-02-03; First posted 2000-02-04 (Estimated); Results first posted 2011-11-22 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-09

CONDITIONS: Abdominal Neoplasm; Colonic Neoplasm; Mesothelioma; Peritoneal Neoplasm
Keywords: Surgery; Mesothelioma; Pseudomyxoma; Colon Cancer; Chemotherapy
MeSH Terms: conditions — Abdominal Neoplasms; Colonic Neoplasms; Mesothelioma; Peritoneal Neoplasms | interventions — Surgical Procedures, Operative; Cytoreduction Surgical Procedures; Cisplatin; Paclitaxel; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Peritoneal mesothelioma (Experimental): Patients with peritoneal mesothelioma suffer with intractable ascites but have a very surface oriented tumor which usually does not invade into organs and cause organ dysfunction. The main source of symptoms and cause of death is intractable ascites.
  Interventions: Procedure: Surgery; Procedure: Continuous hyperthermic peritoneal perfusion (CHPP) with Cisplatin; Drug: Postoperative dwell with paclitaxel and 5-FU
- Low grade mucinous adenocarcinoma (Experimental): Low grade mucinous adenocarcinoma also includes low grade mucinous neoplasms of borderline malignant potential. Patients with low grade mucinous adenocarcinoma can have prolonged survival with debulking surgery alone. The majority of patients with truly malignant disease will die of complications from intraperitoneal progression of tumor within 2 to 5 years. The tumors are often surface oriented within the peritoneal cavity without metastases to other distant sites. The most common origin for this type of tumor is the appendix and ovary.
  Interventions: Procedure: Surgery; Procedure: Continuous hyperthermic peritoneal perfusion (CHPP) with Cisplatin; Drug: Postoperative dwell with paclitaxel and 5-FU
- Adenocarcinoma of gastrointestinal origin (Experimental): Adenocarcinoma of gastrointestinal origin also includes other than low grade mucinous. Aggressive gastrointestinal adenocarcinomas such as gastric, small bowel, and colon cancer , tend to be more invasive into tissues and can more readily metastasize to distant sites. The cause of death is usually directly related to intraperitoneal progression of tumor. It is a more difficult group of patients to treat with intraperitoneal therapy because of the aggressive and invasive nature of the tumors.
  Interventions: Procedure: Surgery; Procedure: Continuous hyperthermic peritoneal perfusion (CHPP) with Cisplatin; Drug: Postoperative dwell with paclitaxel and 5-FU

INTERVENTIONS:
Procedure: Surgery — Patients will undergo cytoreductive surgery to remove as much tumor as possible. Part of the intestines, pancreas, stomach or the entire spleen may also be removed if they are affected.
  Other Names: Cytoreductive surgery
Procedure: Continuous hyperthermic peritoneal perfusion (CHPP) with Cisplatin
  Other Names: Platinol; Cisplatinum
Drug: Postoperative dwell with paclitaxel and 5-FU — Intraperitoneal dwell chemotherapy with a combination of 5-FU and Paclitaxel will be delivered in the early postoperative period (day 7 today 12 after surgery). Patients will be premedicated with hydrocortisone (100 mg/intravenous push (i.v.p.)), diphenhydramine (50 mg i.v.p.) and ranitidine (50 mg i.v.p.) 30 minutes prior to delivering intraperitoneal chemotherapy. One liter of normal saline will be infused containing 5-FU (800 mg/M^2) and 1 L of normal saline containing paclitaxel (125 mg/M^2) will be infused over 60 minutes. The chemotherapy solution will be left in the abdominal cavity permanently for slow absorption.
  Other Names: 5-FU

SUMMARY:
This study will test the effectiveness of an experimental treatment for peritoneal cancer involving surgical removal of the tumor, perfusion of the abdomen during surgery with a heated solution of the drug cisplatin, and post-surgery combination chemotherapy in the abdomen with fluorouracil (5-FU) and paclitaxel.

Patients with certain peritoneal cancer whose tumors are confined to the abdomen may be eligible for this study. Candidates are screened with a medical history and physical examination, including blood tests, electrocardiogram and possibly bone scan, brain magnetic resonance imaging (MRI), and chest, abdomen and pelvic CT scans.

Participants undergo surgery to remove as much tumor as possible. Part of the intestines, pancreas, stomach or the entire spleen may also be removed if they are affected. During surgery, after the tumor has been removed, two catheters (thin plastic tubes) are placed in the abdomen. A chemotherapy solution containing the anti-cancer drug cisplatin heated to a temperature of about 108.6 degrees (10 degrees above normal body temperature) is then delivered into the abdomen through one catheter and drained through another. During treatment, a drug called sodium thiosulfate is given through a vein to reduce the risk of side effects of cisplatin, particularly kidney damage. After 90 minutes of bathing the abdomen with this solution, the drug is rinsed from the abdomen and the catheters removed. Another small catheter is then placed and left inside the abdomen with one end coming out through the skin. Seven to 12 days after the operation, the anti-cancer drugs 5-FU and paclitaxel are given through this catheter.

After complete recovery from the surgery, the catheter is removed and the patient is discharged from the hospital. Clinic visits are scheduled for periodic follow-up examination, imaging, and tests 3 and 6 months after surgery and every 6 months for up to 5 years as long as the disease does not worsen. Patients whose disease progresses are taken off the study and referred back to their local physician or referred for alternative care or other research studies.

Patients are also asked to assess how this therapy affects their general health and well being. This will require filling out two quality-of-life (QOL) questionnaires before surgery and again at each follow-up visit after surgery. Each questionnaire takes about 15 minutes to complete.

DETAILED DESCRIPTION:
Background:

Cytoreductive surgery plus aggressive combination intraperitoneal chemotherapy may significantly alter the natural history of peritoneal carcinomatosis. The purpose of this study is to examine the treatment results of continuous hyperthermic peritoneal perfusion (CHPP) with cisplatin plus early postoperative intraperitoneal dwell therapy with 5-FU and paclitaxel after cytoreductive surgery for peritoneal carcinomatosis.

Objectives:

The primary objective of this study is to determine response and survival after continuous hyperthermic peritoneal perfusion with cisplatin and early postoperative intraperitoneal dwell therapy with 5-FU and paclitaxel. Response can only be assessed by measuring the time to clinical or radiographic recurrence of disease.

The secondary objectives include the determination of pharmacokinetics of paclitaxel and 5-FU delivered into the peritoneal cavity and the impact that continuous hyperthermic peritoneal perfusion with cisplatin and early postoperative intraperitoneal dwell therapy with 5-FU and paclitaxel has on patients' health related quality of life.

The evaluation of pure populations of tumor and normal mesothelial cells to

* determine if signal transduction pathways are distinct in tumor versus normal tissue
* to see if specific cell pathways are activated or inhibited as a consequence of therapy.
* to validate that this technology can provide informative data about these events as a potential surrogate for clinical benefit from therapy or biological behavior of the tumor.

Eligibility:

The patient greater than or equal to 30 kg must have histologically proven peritoneal carcinomatosis from one of the following histologies: 1) primary peritoneal mesothelioma; 2) low grade mucinous adenocarcinoma (including low grade mucinous neoplasms of borderline malignant potential); 3) adenocarcinoma of gastrointestinal tract origin (other than low grade mucinous, excluding pancreatic cancer), with disease confined to the peritoneal cavity. Patients may not have had treatment for their disease within the previous 30 days and have recovered from all toxicity. Patients must meet certain safety laboratory criteria and may not have major medical disorders that would place them at unacceptable risk for a major surgical procedure. Patients may not have received prior intraperitoneal platinum therapy.

Design:

Patients will undergo cytoreductive surgery followed by CHPP with cisplatin. A peritoneal dialysis catheter will be inserted into the peritoneal cavity at the time of laparotomy. In the early postoperative period (day 2 - 10) intraperitoneal dwell chemotherapy with paclitaxel (125 mg/M^2) and 5-FU (800 mg/M^2) will be administered. Patients will be seen 4 - 6 weeks after discharge for a physical examination and laboratory screen and QOL evaluation. Tumor marker will be included at this stage. Patients will then be seen every 3 months for the first year after surgery and every 6 months thereafter. At each visit they will undergo physical examination, laboratory screening (including tumor marker) and a CT scan of the chest, abdomen and pelvis and QOL evaluation.

The objective of this pilot study is to estimate the ability of peritoneal perfusion to achieve potentially tolerable disease free survival in patients with a variety of tumors. For each class of tumors, an appropriate, distinct median disease free survival will be targeted as the principal endpoint. The trial will be conducted as a set of three single-stage phase II studies, with an early stopping rule for clearly unacceptable outcomes. It is expected that accrual for 59 patients with adenocarcinoma of gastrointestinal origin (other than low grade mucinous), 48 patients with low grade mucinous adenocarcinoma, and 96 patients with primary peritoneal mesothelioma (total accrual of 203) will require approximately 5 -6 years.

Results will be assessed by following the time to radiographic or clinical recurrence of disease and survival. Patients will be stratified for entry based on histology. This will include 3 cohorts: 1) peritoneal mesothelioma; 2) low grade mucinous adenocarcinoma (including low grade mucinous neoplasms of borderline malignant potential); and 3) adenocarcinoma of gastrointestinal origin (other than low grade mucinous).

ELIGIBILITY:
* INCLUSION CRITERIA:

The patient must have histologically proven peritoneal carcinomatosis from the following histologies: primary peritoneal mesothelioma; low grade mucinous adenocarcinoma (including low grade mucinous neoplasms of borderline malignant potential); adenocarcinoma of gastrointestinal tract origin (other than low grade mucinous, excluding pancreatic cancer).

Radiologic workup must demonstrate that the disease is confined to the peritoneal cavity.

Radiologic workup or prior abdominal exploration must be consistent with disease which can be debulked to a residual size of less that 1 cm in diameter per tumor deposit.

Patients must have an Eastern Cooperative Onocology Group (ECOG) performance status of less than or equal to 2.

Patients must have a minimum expected duration of survival of greater than 8 weeks.

Patients must have recovered from any toxicity from all prior chemotherapy, immunotherapy or radiotherapy and be at least 30 days past the date of their last treatment.

EXCLUSION CRITERIA:

Patients will be excluded if they have concomitant medical problems that would place them at unacceptable risk for a major surgical procedure.

Patients at increased risk for coronary artery disease or cardiac dysfunction (e.g., age greater than 65, history of hypertension, first degree relative with atherosclerotic coronary artery disease) will undergo cardiac evaluation and will not be eligible if they demonstrate significant irreversible ischemia on a stress thallium study or an injection fraction of less than 40 percent.

Patients who have shortness of breath with minimal exertion and who are at risk for pulmonary disease (e.g., chronic smokers) will undergo pulmonary function testing and will not be eligible if their forced expiratory volume 1 (FEV1) is less than 1.2 liters or their maximum voluntary ventilation is less than 50 percent of expected.

Patients who have a baseline neurological toxicity of Grade 3 or greater will be excluded because of the potential neurotoxicity associated with platinum and paclitaxel therapy.

Patients will be ineligible if they have a creatinine of greater than 1.5 or a creatinine clearance of less 70 mL/min.

Patients will be ineligible if the white blood cell (WBC) is less than 3000/microliters or platelets are less than 75,000mL/mm(3).

Patients must have a serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) within 5 times the upper limit of normal and a total serum bilirubin of less than 3 times the upper limit of normal, both of which define the upper limit of grade 2 treatment related toxicities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2000-01; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marybeth S Hughes, M.D., Principal Investigator — National Cancer Institute, National Institutes of Health
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Dedrick RL, Myers CE, Bungay PM, DeVita VT Jr. Pharmacokinetic rationale for peritoneal drug administration in the treatment of ovarian cancer. Cancer Treat Rep. 1978 Jan;62(1):1-11. PMID 626987
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2000-C-0069.html
- See also: Medline Plus — http://www.nlm.nih.gov/medlineplus/
- See also: Drug Information — http://druginfo.nlm.nih.gov/drugportal/drugportal.jsp
- See also: US FDA Resources — http://www.clinicaltrials.gov/ct2/info/fdalinks

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total accrual of 203 was expected within approximately 5-6 years (59 patients for adenocarcinoma of gastrointestinal origin, other than low grade mucinous; 48 patients with low grade mucinous adenocarcinoma; and 96 patients with primary peritoneal mesothelioma).
Period: Overall Study
Arm/Group | Peritoneal Mesothelioma | Low Grade Mucinous Adenocarcinoma | Adenocarcinoma of Gastrointestinal Origin
Started | 83 | 48 | 57
Not Evaluable | 21 | 9 | 23
Completed | 61 | 39 | 35
Not Completed | 22 | 9 | 22

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Peritoneal Mesothelioma | Low Grade Mucinous Adenocarcinoma | Adenocarcinoma of Gastrointestinal Origin | Total
Number analyzed (Participants) | 83 | 48 | 57 | 188
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 0 | 0 | 3
  Between 18 and 65 years | 71 | 43 | 52 | 166
  >=65 years | 9 | 5 | 5 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.95 (14.12) | 50.48 (10.85) | 49.70 (11.78) | 50.01 (12.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 23 | 28 | 89
  Male | 45 | 25 | 29 | 99
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 69 | 38 | 54 | 161
  Hispanic | 6 | 0 | 3 | 9
  African American | 2 | 7 | 0 | 9
  Asian American | 4 | 3 | 0 | 7
  Unknown | 2 | 0 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 83 | 48 | 57 | 188

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Disease-free Survival
Description: Participants who achieve either a six or twelve month disease free interval based on radiographic imaging and symptoms.
Time Frame: On study date until the first scan with imageable disease, assessed up to 100 months or more.
Population: This outcome measure was not analyzed because information was not consistently available.
Arm/Group | Peritoneal Mesothelioma | Low Grade Mucinous Adenocarcinoma | Adenocarcinoma of Gastrointestinal Origin
Number analyzed (Participants) | 0 | 0 | 0

2. Primary Outcome: Number of Participants With a Response
Description: Response is assessed by measuring the time to clinical or radiographic recurrence of disease. Patients will be followed with computed tomography (CT) scans. At any time point where there is evidence of progressive disease in the peritoneal cavity (imageable tumor nodules or new onset of ascites) the patients will be scored as failing within the abdominal cavity.
Time Frame: Patients were assessed every three months for one year and then every 6 months
Measure: Number; unit: Participants
Arm/Group | Peritoneal Mesothelioma | Low Grade Mucinous Adenocarcinoma | Adenocarcinoma of Gastrointestinal Origin
Number analyzed (Participants) | 83 | 48 | 57
Participants | 24 | 18 | 6

3. Primary Outcome: Number of Participants With Adverse Events
Description: Here are the number of participants with adverse events. For the detailed list of adverse events see the adverse event module.
Time Frame: only assessed during the perioperative period (i.e. up to 90 days following surgery)
Population: 188 participants is consistent with the total number of participants analyzed (e.g. total from each column in participant flow, 83 P. Meso + 48 L. Grade + 57 Adeno. = 188).
Measure: Number; unit: Participants
Groups:
- Mesothelioma, Low Grade, and Adenocarcinoma: Patients with peritoneal mesothelioma suffer with intractable ascites. Patients with low grade mucinous adenocarcinoma can have prolonged survival with debulking surgery alone. Adenocarcinoma of gastrointestinal origin also includes other than low grade mucinous. Aggressive gastrointestinal adenocarcinomas such as gastric, small bowel, and colon cancer, tend to be more invasive.
Arm/Group | Mesothelioma, Low Grade, and Adenocarcinoma
Number analyzed (Participants) | 188
Participants | 73

4. Secondary Outcome: Percentage of Participants Who Had Paclitaxel and 5-fluorouracil (5-FU) Analysis Performed
Description: Paclitaxel and 5-FU levels in plasma and perfusate will be determined by standard high-performance liquid chromatography (HPLC). Samples will be collected just prior to (Time 0) the infusion of the intraperitoneal dwell of 5-FU and paclitaxel, at the following time intervals after the conclusion of the intraperitoneal dwell infusion (15 minutes, 1 hour, 6 hour, 12 hour, 24 hour, 48 hour).
Time Frame: Perioperative day 7-12 after surgery
Population: This outcome measure was not analyzed because it was not feasible (e.g. inadequate samples).
Arm/Group | Peritoneal Mesothelioma | Low Grade Mucinous Adenocarcinoma | Adenocarcinoma of Gastrointestinal Origin
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Quality of Life Questionnaire Score
Description: The Short-Form-36 Health Survey (SF-36) and the Functional Assessment of Cancer Therapy Disease Specific for Colorectal Cancer (FACT-C) will be given to the patients upon admission preoperatively, then 6 weeks postoperatively, and then 3, 6, 9, and 12 months for the first year and then every 6 months until the patient goes off study. These forms summarize a participants positive and negative aspects that characterize one's psychological (emotional(, physical, and social well-being at a point in time.
  For detailed information about the questionnaires, please see the Protocol Link module.
Time Frame: preop, 6 weeks postop and then 3, 6, 9, and 12 months the first year and then every 6 months until the patient is off study
Population: This outcome measure was not evaluated due to poor patient compliance.
Arm/Group | Peritoneal Mesothelioma | Low Grade Mucinous Adenocarcinoma | Adenocarcinoma of Gastrointestinal Origin
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Signal Transduction Pathways in Tumor Tissue Versus Normal Tissue
Description: Signal transduction pathways were measured using reverse phase protein lysate microarray to determine if the pathways are distinct in tumor versus normal tissue.
Time Frame: once during surgery
Population: This outcome measure was not analyzed because it was not feasible.
Groups:
- Normal Tissue: Non-diseased tissue
- Tumor Tissue: Diseased tissue
Arm/Group | Normal Tissue | Tumor Tissue
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: Adverse Events: 188 participants is consistent with the total number of participants analyzed (e.g. total from each column in participant flow, 83 P.Meso + 48 L.Grade + 57 Adeno. = 188).
Arm/Group | Mesothelioma, Low Grade, and Adenocarcinoma
Serious Adverse Events (participants affected / at risk) | 71/188
Other Adverse Events (participants affected / at risk) | 2/188
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mesothelioma, Low Grade, and Adenocarcinoma (N=188)
ascites (Gastrointestinal disorders) | 2 (2)
atrial fibrillation (Cardiac disorders) | 1 (1)
cholecystitis (Hepatobiliary disorders) | 1 (1)
colitis (Gastrointestinal disorders) | 1 (1)
colon perforation (Gastrointestinal disorders) | 2 (2)
diarrhea (Gastrointestinal disorders) | 1 (1)
Deep venous thrombosis (DVT) (Vascular disorders) | 1 (1)
Enterocutaneous fistula (Gastrointestinal disorders) | 2 (2)
Gastric perforation (Gastrointestinal disorders) | 1 (1)
Gastrointestinal (GI) perforation (Gastrointestinal disorders) | 1 (1)
Hallucinations/post operative (op) psychosis (Psychiatric disorders) | 2 (2)
Ileus (Gastrointestinal disorders) | 2 (2)
Myocardial infarction (Cardiac disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (4)
Neutropenic fever (Infections and infestations) | 5 (5)
Pancreatic fistula (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 3 (3)
Pulmonary embolism (PE) (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pelvic abscess (Reproductive system and breast disorders) | 1 (1)
Perforated bowel (Gastrointestinal disorders) | 1 (1)
Peritonitis (Gastrointestinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 2 (2)
Small bowel obstruction (sbo) (Gastrointestinal disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Small bowel obstruction (Gastrointestinal disorders) | 12 (12)
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thrombosis jugular (Vascular disorders) | 1 (1)
Thrombosis portal vein (Hepatobiliary disorders) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 1 (1)
Voice changes (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wound infection (Infections and infestations) | 7 (7)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mesothelioma, Low Grade, and Adenocarcinoma (N=188)
Sinus ventricular tachycardia (SVT) (Cardiac disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No